CLINICAL TRIAL: NCT06411665
Title: Effect of Oliceridine Analgesia on Postoperative Nause and Vomiting in Laparoscopic Colorectal Surgery: A Randomized Trial
Brief Title: Effect of Oliceridine Analgesia on Postoperative Nause and Vomiting
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Chairman of Department of Anesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024-073
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperative nausea and vomiting; Laparoscopic colorectal surgery; Postoperative analgesia; Oliceridine
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine; Injections; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oliceridine group (Experimental): Patient-controlled analgesia pump is provided immediately after surgery. The pump is established with oliceridine 15 mg, diluted with normal saline to 100 ml, and programmed to deliver 2-ml boluses with a 10-min lockout interval and a background infusion rate at 1 ml/h. The pump will be used during the first 3 days after surgery.
  Interventions: Drug: Oliceridine
- Morphine group (Active Comparator): Patient-controlled analgesia pump is provided immediately after surgery. The pump is established with morphine 50 mg, diluted with normal saline to 100 ml, and programmed to deliver 2-ml boluses with a 10-min lockout interval and a background infusion rate at 1 ml/h. The pump will be used during the first 3 days after surgery.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Oliceridine — Patient-controlled intravenous analgesia with oliceridine for up to 3 days after surgery.
  Other Names: Oliceridine for injection
  Arms: Oliceridine group
Drug: Morphine — Patient-controlled intravenous analgesia with morphine for up to 3 days after surgery.
  Other Names: Morphine for injection
  Arms: Morphine group

SUMMARY:
Postoperative nausea and vomiting (PONV) is common after surgery and impede rapid recovery after surgery. Patients who undergo laparoscopic colorectal surgery are more likely to develop PONV due to the pneumoperitoneum, interruption of gastrointestinal system, delay of oral feeding, and nasogastric catheterization, as well as postoperative opioid analgesic requirement to control acute pain. Oliceridine is a novel selective μ-opioid agonist. It stimulates G protein signalling but is markedly less potent than morphine for β-arrestin recruitment; the latter contributes to opioid-related adverse events including PONV. It is postulated that G protein-biased agonists may deliver effective analgesia with fewer opioid-related adverse events. This randomized trial aimed to investigate whether oliceridine for patient-controlled analgesia can decrease the incidence of PONV in patients recovering from laparoscopic colorectal surgery.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is a common adverse event after surgery. A retrospective study found that PONV occurred in 14.4% of enrolled 106860 patients. The reported incidences in prospective studies varied between 25.5% to 33.3%. Certain types of laparoscopic surgery are associated with an increased risk of PONV, including bariatric surgery, gynecological surgery, and cholecystectomy. PONV can lead to dehydration and electrolyte imbalances, delay early ambulation, impede rapid recovery after surgery, decrease patients' satisfactory, and potentially prolong hospital stay and increase cost.

Opioids are commonly used during the perioperative period and are associated with increased PONV. Conventional opioids such as morphine and sufentanil activate both the G protein and β-arrestin pathways; the latter approach contributes to opioid-related PONV through multiple mechanisms, such as enhanced vestibular sensitivity, direct effects on the chemoreceptor trigger zone, and delayed gastric emptying. Oliceridine is a novel selective μ-opioid agonist. It stimulates G protein signalling but is markedly less potent than morphine for β-arrestin recruitment. It is therefore postulated that G protein-biased agonists may deliver effective analgesia with fewer opioid-related PONV.

Previous studies in patients with moderate-to-severe pain following orthopaedic surgery-bunionectomy or plastic surgery-abdominoplasty showed that oliceridine provided an excellent analgesic efficacy compared with morphine and placebo. The analgesic efficiency of 0.35 mg or 0.5 mg oliceridine was equal to 1 mg morphine. However, the rate of PONV was significantly lower in patients given oliceridine than in those given morphine. Patients who undergo laparoscopic colorectal surgery are more likely to develop PONV due to the pneumoperitoneum, interruption of gastrointestinal system, delay of oral feeding, and nasogastric catheterization, as well as postoperative opioid analgesia to control pain. Thus, selective μ-opioid agonist might be more suitable for postoperative analgesia for these patients.

This randomized trial aimed to investigate whether oliceridine compared with morphine for postoperative analgesia can decrease the incidence of PONV in patients after laparoscopic colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 80 years;
2. Scheduled to undergo elective laparoscopic colorectal surgery;
3. Required patient-controlled intravenous analgesia.

Exclusion Criteria:

1. Pregnancy.
2. Severe heart dysfunction (New York Heart Association functional classification 4), hepatic insufficiency (Child-Pugh grade C), renal insufficiency (serum creatinine of 442 μmol/L or above, or requirement of renal replacement therapy), or Amercian Society of Anesthesiologists classification IV or above.
3. Unable to complete preoperative assessment due to severe dementia or language barrier.
4. Other conditions that are considered unsuitable for study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative nause and vomiting (PONV) with 72 hours. | Up to 72 hours after surgery.
  Defined as the development of any nausea, retching, or vomiting within 72 h after surgery.

SECONDARY OUTCOMES:
The incidence of postoperative vomiting within 72 hours. | Up to 72 hours after surgery
  Defined as the development of any retching or vomiting within 72 h after surgery.
Area under curve of nausea intensity at predefined timepoints. | Up to 72 hours after surgery
  Nausea intensity is assessed with the numeric rating scale, an 11-point scale where 0=no nausea and 10=the most severe nausea.
Area under curve of pain intensity at rest at predefined timepoints. | Up to 72 hours after surgery
  Pain intensity is assessed with the numeric rating scale, an 11-point scale where 0=no pain and 10=the worst pain.
Area under curve of pain intensity with movement at predefined timepoints | Up to 72 hours after surgery
  Pain intensity is assessed with the numeric rating scale, an 11-point scale where 0=no pain and 10=the worst pain.
Quality of recovery at 24 hours and 72 hours after surgery. | Up to 72 hours after surgery
  Quality of recovery (QoR) is assessed with the QOR-15 scale, a 15-item scale that provides a global measure of postoperative recovery, with a score ranging from 0 (extremely poor QoR) to 150 (excellent QoR).
Time to first flatus after surgery. | Up to 5 days after surgery.
  Time to first flatus after surgery.

OTHER OUTCOMES:
Time to first ambulation after surgery. | Up to 5 days after surgery.
  Time to first ambulation after surgery.
Patients' satisfaction score with postoperative analgesia. | At 72 hours after surgery.
  Patients' satisfaction is assessed with a visual analogue scale, a 0-100 scale where 0=very dissatisfied and 100=very satisfied.
Total opioid consumption within 72 hours after surgery. | Up to 72 hours after surgery.
  Total opioid consumption within 72 hours after surgery.
Subjective sleep quality during the first 3 nights after surgery. | Up to 72 hours after surgery.
  Subjective sleep quality is assessed with the numeric rating scale, an 11-point scale where 0=the best sleep and 10=the worst sleep.
Length of hospital stay after surgery. | Up to 30 days after surgery.
  Length of hospital stay after surgery.
Major complications within 30 days after surgery. | Up to 30 days after surgery.
  Major complications are defined as new-onset medical events that are deemed harmful and required therapeutic intervention, that is grade II or higher on the Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, PHD, Study Director — Peking University First Hospital
Locations (1):
- Dong-Xin Wang, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim JH, Cheon BR, Kim MG, Hwang SM, Lim SY, Lee JJ, Kwon YS. Postoperative Nausea and Vomiting Prediction: Machine Learning Insights from a Comprehensive Analysis of Perioperative Data. Bioengineering (Basel). 2023 Oct 1;10(10):1152. doi: 10.3390/bioengineering10101152. PMID 37892882
- [Result] Matsumoto A, Satomi S, Kakuta N, Narasaki S, Toyota Y, Miyoshi H, Horikawa YT, Saeki N, Tanaka K, Tsutsumi YM. Remimazolam's Effects on Postoperative Nausea and Vomiting Are Similar to Those of Propofol after Laparoscopic Gynecological Surgery: A Randomized Controlled Trial. J Clin Med. 2023 Aug 20;12(16):5402. doi: 10.3390/jcm12165402. PMID 37629444
- [Result] DREAMS Trial Collaborators and West Midlands Research Collaborative. Dexamethasone versus standard treatment for postoperative nausea and vomiting in gastrointestinal surgery: randomised controlled trial (DREAMS Trial). BMJ. 2017 Apr 18;357:j1455. doi: 10.1136/bmj.j1455. PMID 28420629
- [Result] Song Y, Zhu J, Dong Z, Wang C, Xiao J, Yang W. Incidence and risk factors of postoperative nausea and vomiting following laparoscopic sleeve gastrectomy and its relationship with Helicobacter pylori: A propensity score matching analysis. Front Endocrinol (Lausanne). 2023 Feb 22;14:1102017. doi: 10.3389/fendo.2023.1102017. eCollection 2023. PMID 36909334
- [Result] Myles PS, Williams DL, Hendrata M, Anderson H, Weeks AM. Patient satisfaction after anaesthesia and surgery: results of a prospective survey of 10,811 patients. Br J Anaesth. 2000 Jan;84(1):6-10. doi: 10.1093/oxfordjournals.bja.a013383. PMID 10740539
- [Result] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Result] Suh S, Helm M, Kindel TL, Goldblatt MI, Gould JC, Higgins RM. The impact of nausea on post-operative outcomes in bariatric surgery patients. Surg Endosc. 2020 Jul;34(7):3085-3091. doi: 10.1007/s00464-019-07058-5. Epub 2019 Aug 6. PMID 31388805
- [Result] Habib AS, Chen YT, Taguchi A, Hu XH, Gan TJ. Postoperative nausea and vomiting following inpatient surgeries in a teaching hospital: a retrospective database analysis. Curr Med Res Opin. 2006 Jun;22(6):1093-9. doi: 10.1185/030079906X104830. PMID 16846542
- [Result] Gan TJ, Belani KG, Bergese S, Chung F, Diemunsch P, Habib AS, Jin Z, Kovac AL, Meyer TA, Urman RD, Apfel CC, Ayad S, Beagley L, Candiotti K, Englesakis M, Hedrick TL, Kranke P, Lee S, Lipman D, Minkowitz HS, Morton J, Philip BK. Fourth Consensus Guidelines for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2020 Aug;131(2):411-448. doi: 10.1213/ANE.0000000000004833. PMID 32467512
- [Result] Mauermann E, Clamer D, Ruppen W, Bandschapp O. Association between intra-operative fentanyl dosing and postoperative nausea/vomiting and pain: A prospective cohort study. Eur J Anaesthesiol. 2019 Nov;36(11):871-880. doi: 10.1097/EJA.0000000000001081. PMID 31567573
- [Result] Zhang R, Zhang WX, Ma XR, Feng Y. Intraoperative Sufentanil Consumption and the Risk of Postoperative Nausea and/or Vomiting: A Retrospective Observational Study. Pain Ther. 2023 Oct;12(5):1271-1281. doi: 10.1007/s40122-023-00546-6. Epub 2023 Aug 9. PMID 37556070
- [Result] Smith HS, Laufer A. Opioid induced nausea and vomiting. Eur J Pharmacol. 2014 Jan 5;722:67-78. doi: 10.1016/j.ejphar.2013.09.074. Epub 2013 Oct 21. PMID 24157979
- [Result] DeWire SM, Yamashita DS, Rominger DH, Liu G, Cowan CL, Graczyk TM, Chen XT, Pitis PM, Gotchev D, Yuan C, Koblish M, Lark MW, Violin JD. A G protein-biased ligand at the mu-opioid receptor is potently analgesic with reduced gastrointestinal and respiratory dysfunction compared with morphine. J Pharmacol Exp Ther. 2013 Mar;344(3):708-17. doi: 10.1124/jpet.112.201616. Epub 2013 Jan 8. PMID 23300227
- [Result] Markham A. Oliceridine: First Approval. Drugs. 2020 Nov;80(16):1739-1744. doi: 10.1007/s40265-020-01414-9. PMID 33025536
- [Result] Singla NK, Skobieranda F, Soergel DG, Salamea M, Burt DA, Demitrack MA, Viscusi ER. APOLLO-2: A Randomized, Placebo and Active-Controlled Phase III Study Investigating Oliceridine (TRV130), a G Protein-Biased Ligand at the mu-Opioid Receptor, for Management of Moderate to Severe Acute Pain Following Abdominoplasty. Pain Pract. 2019 Sep;19(7):715-731. doi: 10.1111/papr.12801. Epub 2019 Jun 24. PMID 31162798
- [Result] Viscusi ER, Skobieranda F, Soergel DG, Cook E, Burt DA, Singla N. APOLLO-1: a randomized placebo and active-controlled phase III study investigating oliceridine (TRV130), a G protein-biased ligand at the micro-opioid receptor, for management of moderate-to-severe acute pain following bunionectomy. J Pain Res. 2019 Mar 11;12:927-943. doi: 10.2147/JPR.S171013. eCollection 2019. PMID 30881102
- [Result] Hammer GB, Khanna AK, Michalsky C, Wase L, Demitrack MA, Little R, Fossler MJ, Ayad S. Oliceridine Exhibits Improved Tolerability Compared to Morphine at Equianalgesic Conditions: Exploratory Analysis from Two Phase 3 Randomized Placebo and Active Controlled Trials. Pain Ther. 2021 Dec;10(2):1343-1353. doi: 10.1007/s40122-021-00299-0. Epub 2021 Aug 5. PMID 34351590
- [Result] Beard TL, Michalsky C, Candiotti KA, Rider P, Wase L, Habib AS, Demitrack MA, Fossler MJ, Viscusi ER. Oliceridine is Associated with Reduced Risk of Vomiting and Need for Rescue Antiemetics Compared to Morphine: Exploratory Analysis from Two Phase 3 Randomized Placebo and Active Controlled Trials. Pain Ther. 2021 Jun;10(1):401-413. doi: 10.1007/s40122-020-00216-x. Epub 2020 Nov 18. PMID 33210266
- [Result] Liu Y, Xiao S, Yang H, Lv X, Hou A, Ma Y, Jiang Y, Duan C, Mi W; CAPOPS Group. Postoperative pain-related outcomes and perioperative pain management in China: a population-based study. Lancet Reg Health West Pac. 2023 Jun 10;39:100822. doi: 10.1016/j.lanwpc.2023.100822. eCollection 2023 Oct. PMID 37927993